CLINICAL TRIAL: NCT02383147
Title: A Monocentric Study for Development and Use of Tomographic Neurofeedback Protocols for Patients Suffering From Chronic Tinnitus
Brief Title: Efficacy Study for Development and Use of Neurofeedback-trainings for Patients Suffering From Chronic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USZ-ORL-KT-001
Record Dates: First submitted 2015-02-18; First posted 2015-03-09 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Tinnitus, Subjective
Keywords: Adult; Aged; Alpha Rhythm; Auditory Cortex; Chronic; Electroencephalography; Female; Humans; Male; Neurofeedback; Prospective Studies; Questionnaires; Tinnitus; Treatment Outcome
MeSH Terms: conditions — Tinnitus; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Tomographic Neurofeedback (TONF) (Experimental): 15x Neurofeedback Trainings, 1-2 times per week
  Interventions: Device: Tomographic Neurofeedback
- Non Tomographic Neurofeedback (NTE) (Active Comparator): 15x Neurofeedback Trainings, 1-2 times per week
  Interventions: Device: Non Tomographic Neurofeedback

INTERVENTIONS:
Device: Tomographic Neurofeedback — EEG-Electrodes are placed on the patients head to record the brain activity, EEG-recordings are processed by the standardized Low Resolution Brain Electromagnetic Tomography algorithm (sLORETA) to calculate the frequency spectrum in the auditory cortex and deliver feedback for the patient
  Arms: Tomographic Neurofeedback (TONF)
Device: Non Tomographic Neurofeedback — EEG-electrodes are placed on the patients head, but only 4 electrodes (Fc1, Fc2, F3 and F4 of a 10-10 EEG-system) record the surface activity and generate the feedback for the patient.
  Arms: Non Tomographic Neurofeedback (NTE)

SUMMARY:
Chronic tinnitus affects about 10-15% of the population in industrialized countries. Investigations of the brain activity by using electroencephalography (EEG) showed that in localized regions of the hearing system brain activity was decreased. This reduction of activity is thought to be one of the reasons that keep the perception of the tinnitus going. Recent studies have shown that neurofeedback is a viable option for treatment of chronic tinnitus. By using neurofeedback it is possible to train brain functions by the simple principle of rewarding wanted changes and punishing unwanted ones. The purpose of the investigators study is to show the efficacy of specific localized neurofeedback training in comparison to global relaxing neurofeedback training. In order to achieve decreased tinnitus symptoms or even disappearance of the tinnitus, 15 neurofeedback trainings are planned. Before and up to 6 month after the training EEG-recordings are performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Chronic Tinnitus > 0.5 years
* Informed Consent
* Fluent in German language

Exclusion Criteria:

* Psychological and neurological disorders other than tinnitus
* Drug- or Alcohol abuse
* Tranquilizer, antiepileptic drugs, antipsychotics or anesthetics intake
* Impairing hearing loss or Cochlea Implant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-03; Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Tinnitus symptoms assessed by questionnaires | at 1, 3, 6 month follow up
  Assessement of the Tinnitus symptoms before and after the Treatment with neurofeedback by different questionnaires tailored for Tinnitus and Quality of life.
Change from Baseline in delta (3-4Hz) and alpha (8-12Hz) frequency band EEG-activity in the auditory cortex | at 1, 3, 6 month follow up
  EEG recordings of the trained frequency bands are compared before and after the Intervention in the named time periods

SECONDARY OUTCOMES:
Difference in efficacy between Tomographic Neurofeedback (TONF) and Non Tomographic Neurofeedback (NTE) in treatment of tinnitus assessed by tinnitus questionnaires and frequency band EEG-activity measurements (3-4Hz and 8-12Hz) compared to Baseline. | at 1, 3, 6 month follow up
  Investigation if there is a significant benefit in the TONF Group, compared to the non tomographic Group.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kleinjung, Principal Investigator — ENT-Department, University Hospital Zurich
Locations (1):
- University Hospital Zurich, Division of Otorhinolaryngology ORL, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dohrmann K, Weisz N, Schlee W, Hartmann T, Elbert T. Neurofeedback for treating tinnitus. Prog Brain Res. 2007;166:473-85. doi: 10.1016/S0079-6123(07)66046-4. PMID 17956812
- [Background] Crocetti A, Forti S, Del Bo L. Neurofeedback for subjective tinnitus patients. Auris Nasus Larynx. 2011 Dec;38(6):735-8. doi: 10.1016/j.anl.2011.02.003. Epub 2011 May 17. PMID 21592701
- [Background] Hartmann T, Lorenz I, Muller N, Langguth B, Weisz N. The effects of neurofeedback on oscillatory processes related to tinnitus. Brain Topogr. 2014 Jan;27(1):149-57. doi: 10.1007/s10548-013-0295-9. Epub 2013 May 23. PMID 23700271
- [Derived] Riha C, Guntensperger D, Oschwald J, Kleinjung T, Meyer M. Application of Latent Growth Curve modeling to predict individual trajectories during neurofeedback treatment for tinnitus. Prog Brain Res. 2021;263:109-136. doi: 10.1016/bs.pbr.2021.04.013. Epub 2021 May 20. PMID 34243885
- [Derived] Guntensperger D, Thuring C, Kleinjung T, Neff P, Meyer M. Investigating the Efficacy of an Individualized Alpha/Delta Neurofeedback Protocol in the Treatment of Chronic Tinnitus. Neural Plast. 2019 Mar 26;2019:3540898. doi: 10.1155/2019/3540898. eCollection 2019. PMID 31049052